CLINICAL TRIAL: NCT01473199
Title: Multi-centre, Open Label, Prospective, Consecutive Series Registry Database of BioPoly RS Partial Resurfacing Knee Implant
Brief Title: BioPoly RS Knee Registry Study for Cartilage Defect Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioPoly LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1151001
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cartilage Injury; Defect of Articular Cartilage; Cartilage Damage
Keywords: focal defect; focal lesion; chondral lesion; osteochondral lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioPoly RS Implant (Experimental): BioPoly RS Implant
  Interventions: Device: BioPoly RS Partial Resurfacing Knee Implant

INTERVENTIONS:
Device: BioPoly RS Partial Resurfacing Knee Implant — A long term, surgically invasive device for replacement of focal osteochondral defects in the weight bearing region of the femoral condyles.

SUMMARY:
Information will be collected on the pre-op and post-op clinical status of patients with focal cartilage defects of the femoral condyles treated with the BioPoly RS Partial Resurfacing Knee Implant, a permanent orthopaedic implant. The overall aim of the study is to increase the knowledge of patient outcomes such as pain, knee function, level of activity, and overall quality of life after treatment with the device.

DETAILED DESCRIPTION:
Information will be collected on the pre-op and post-op clinical status of patients with focal cartilage defects of the femoral condyles treated with the BioPoly RS Partial Resurfacing Knee Implant, a permanent orthopaedic implant. The overall aim of the study is to increase the knowledge of patient outcomes such as pain, knee function, level of activity, and overall quality of life after treatment with the device. Patients will be followed for 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cartilage lesion located in weight bearing region of medial or lateral femoral condyles that have failed prior therapy (conservative or surgical)
* Lesion classified as ICRS Grade 2, 3, or 4

Exclusion Criteria:

* Body mass index (BMI) of 30 or more
* Osteoarthritis or rheumatoid arthritis
* Gout
* Uncorrected mal-alignment, ligamentous instability, or meniscal tear
* Total meniscectomy
* Kissing lesion on tibia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 months
  Knee function assessment
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 years
  Knee function assessment

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Through 5 years
  Knee function assessment
VAS Pain | Through 5 years
  Visual analogue scale for assessment of pain
Tegner Activity | Through 5 years
  Measurement of patient's activity level
SF-36 | Through 5 years
  Assessment of patient's overall quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Bobic, MD, Study Chair — Nuffield Health, The Grosvenor Hospital Chester; Dinesh Nathwani, MD, Principal Investigator — The London Clinic; Michael McNicholas, MD, Principal Investigator — Aintree University Hospital; Alister Hart, MD, Principal Investigator — Royal National Orthopaedic Hospital
Locations (5):
- United Kingdom (5):
  - Chester Knee Clinic, Nuffield Health The Grosvenor Hospital Chester, Chester, England
  - Aintree University Hospital, Liverpool, England
  - The London Clinic, London, England
  - Charing Cross Hospital, London, England
  - Royal National Orthopaedic Hospital, Stanmore, England

REFERENCES:
- [Result] Nathwani D, McNicholas M, Hart A, Miles J, Bobic V. Partial Resurfacing of the Knee with the BioPoly Implant: Interim Report at 2 Years. JB JS Open Access. 2017 Apr 6;2(2):e0011. doi: 10.2106/JBJS.OA.16.00011. eCollection 2017 Jun 26. PMID 30229214